CLINICAL TRIAL: NCT00208507
Title: Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup Prosthesis Study (28mm)
Brief Title: 28 mm Ceramic-on-Ceramic Acetabular Cup Total Hip Replacement Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COC 28 mm
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2011-02-16 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Joint Diseases
Keywords: Joint Diseases; Non-Inflammatory Degenerative Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delta Ceramax Ceramic-on-Ceramic Acetabular Cup System (Active Comparator): Total hip replacement with a 28 mm ceramic head and liner.
  Interventions: Device: 28 mm ceramic head on ceramic acetabular liner.
- Pinnacle™ Acetabular Cup with Marathon® Polyethylene (Active Comparator): Total hip replacement with 28 mm ceramic head with a polyethylene liner.
  Interventions: Device: 28 mm ceramic head on polyethylene liner

INTERVENTIONS:
Device: 28 mm ceramic head on ceramic acetabular liner. — Total hip replacement with 28 mm ceramic head on ceramic liner articulation
  Other Names: Delta Ceramax™ 28 mm Ceramic-on-Ceramic Acetabular Cup
  Arms: Delta Ceramax Ceramic-on-Ceramic Acetabular Cup System
Device: 28 mm ceramic head on polyethylene liner — Total hip replacement with 28 mm ceramic head on a polyethylene liner articulation.
  Other Names: Detla Ceramax 28 mm ceramic femoral head and Marathon polyethylene liner.
  Arms: Pinnacle™ Acetabular Cup with Marathon® Polyethylene

SUMMARY:
The study is designed to evaluate artificial hips with a 28 mm ceramic head and a ceramic liner to determine whether they perform as well as artificial hips with a 28 mm ceramic head and a polyethylene liner.

DETAILED DESCRIPTION:
Total Hip Arthroplasty (THA) is the surgical reconstruction of the hip joint through replacement of the femoral head and the acetabular articulating surfaces with fixed prosthetic devices. The goals of THA are relief from pain, restoration of function, and correction of deformity. THA is one of the most common adult reconstructive procedures. Over the past 25 years, patients who have needed to have their hip joint replaced, either due to trauma or arthritic disease, typically have had their hip joint bone articular surfaces replaced with a metal hip stem, metal ball head (either stainless steel or chrome cobalt) and a plastic acetabular cup (metal/metal/plastic). While the basic device has remained essentially unchanged over that period, technological advancements in implant designs and materials, and improvements in surgical technique and instrumentation have made THA one of the most durable and successful procedures in medicine. Reproducible, high-quality, short-term and mid-term results are attained regularly, and total hip replacements commonly last 10 to 15 years and longer. The success of this procedure has allowed its expansion into a wider, and often younger and more active population.

In spite of the improvements in THA, little change has occurred for the acetabular cup liner, which is usually made out of Ultra High Molecular Weight Polyethylene plastic (UHMWPe). Because it is plastic and inherently soft and somewhat pliable under load, the cup's articular surface must inevitability wear and produce debris. This biologic response is now thought to be a significant contributor to prosthetic component loosening, a primary failure mode of THR. UHMWPe also degrades with time in the body. As concerns about polyethylene wear and the associated untoward effects of the generated wear debris, and as THA continues to be used in younger and higher-demand patients with increasing life expectancies, interest in ceramic on ceramic total hip prosthesis has been renewed.

An alumina ceramic-on-ceramic acetabular coupling has been employed as an alternative to metal/polyethylene couplings. This ceramic-on-ceramic coupling has many advantages, including the elimination of polyethylene from the device system, wear rates that are appreciably less than those experienced with metal/polyethylene couplings and reduced biologic reactivity. The potential benefits of an alumina ceramic/ceramic bearing are significant.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease. Composite diagnoses of NIDJD include osteoarthritis, avascular necrosis, post-traumatic arthritis, slipped capital femoral epiphysis (SCFE), fracture of the pelvis, and developmental dysplasia.
* X-ray evaluation confirms the presence of NIDJD
* Femoral and acetabular bone stock is sufficient, regarding strength and shape, and is suitable to receive the implants.
* Individuals 20 to 75 years of age at the time of surgery
* Patients with a previous total hip replacement of the contralateral leg who have a pain rating of none or slight and who are at least one year post arthroplasty are eligible for participation in the study.
* Harris Hip Score of 70 or lower
* Pain at least Moderate

Exclusion Criteria:

* Presence of a previous prosthetic hip replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) in the hip joint to be operated.
* Previous Girdlestone procedure (resection arthroplasty) or surgical fusion of the hip to be operated.
* Acute femoral neck fracture.
* Above knee amputation of the contralateral and/or ipsilateral leg.
* Patients with bilateral degenerative joint disease requiring staged or simultaneous hip replacements.
* Patients with an existing total hip arthroplasty in the contralateral hip with a Harris Hip pain rating of mild, moderate, marked or totally disabled.
* Patients who have undergone total hip arthroplasties in their contralateral hips within the past 12 months.
* Patients with a known allergy to metal (e.g. jewelry).
* Skeletally immature patients (tibial and femoral epiphyses are not closed). Evidence of active infections that may spread to other areas of the body (e.g., osteomyelitis, pyogenic infection of the hip joint, overt infection, urinary tract infection, etc.).
* The presence of highly communicable disease or diseases that may limit follow-up (e.g., immuno-compromised conditions, hepatitis, active tuberculosis, etc.).
* Presence of known metastatic or neoplastic disease.
* Significant neurologic or musculoskeletal disorders or disease that may adversely affect gait or weight bearing, (e.g., muscular dystrophy, multiple sclerosis).
* Conditions that may interfere with the total hip arthroplasty's survival or outcome, (e.g., Paget's disease, Charcot's disease).
* Any patient believed to be unwilling or unable to comply with a rehabilitation program for a cementless total hip replacement or who indicates difficulty or inability to return for follow-up visits prescribed by the study protocol.
* Patient is known to be pregnant, a prisoner, mentally incompetent, and/or alcohol or drug abuser.
* Any systemic steroid therapy, excluding inhalers, within three months prior to surgery.
* Patients carrying the diagnosis of inflammatory degenerative arthritis (IDJD) to include the following composite diagnoses: rheumatoid arthritis, systemic lupus erythematosus, pigmented villonodular synovitis, juvenile rheumatory arthritis and other arthritic processes of inflammatory or autoimmune etiology.
* Patients requiring structural bone grafts in order to support the prosthetic component(s) or to shape the bone to receive the implant(s).
* Patients who refuse to provide consent to participate in the clinical investigation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2003-04-01 (Actual); Primary Completion 2012-01-05 (Actual); Study Completion 2012-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Politi, MD, Principal Investigator — Cardinal Orthopaedic Institute; Douglas Dennis, MD, Principal Investigator — Colorado Joint Replacement
Locations (2):
- United States (2):
  - Colorado Joint Replacement, Denver, Colorado
  - Cardinal Orthopaedic Institute, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected for recruitment into the study from the general diagnosis population defined as "primary total hip arthroplasty (THA) for non-inflammatory degenerative joint disease (NIDJD)." The investigation was conducted at 8 centers. Each center randomly assigned patients to both the investigational and control treatment groups.
Groups:
- Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System: The Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup Prosthesis System consists of a modular ceramic bearing insert that attaches to a Pinnacle™ Acetabular Shell by a taper locking mechanism. The ceramic insert is designed to articulate against a 28 mm ceramic femoral head that is attached to a conventional femoral stem to complete the total hip prosthesis.
- Pinnacle™ Acetabular Cup With Marathon® Polyethylene: Pinnacle™ acetabular shells are a hemispherical type of acetabulum replacement prosthesis that incorporates Porocoat® porous coating for biologic fixation to host bone. The 28mm ceramic femoral heads were used with Marathon® polyethylene liners. The polyethylene insert is designed to articulate against a 28 mm ceramic femoral head that is attached to a conventional femoral stem to complete the total hip prosthesis.
Period: Overall Study
Arm/Group | Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System | Pinnacle™ Acetabular Cup With Marathon® Polyethylene
Started | 177 | 87
Completed | 163 | 79
Not Completed | 14 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System | Pinnacle™ Acetabular Cup With Marathon® Polyethylene | Total
Number analyzed (Participants) | 177 | 87 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.6) | 57.3 (10.3) | 56.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 40 | 127
  Male | 90 | 47 | 137
Region of Enrollment [Count of Participants; unit: Participants]
  United States: United States | 177 | 87 | 264

OUTCOME MEASURES:

1. Primary Outcome: Harris Hip Total Score
Description: The Harris Hip scoring system assigns a numeric value to responses from patients and assessments made by a surgeon. Scores ranges from a minimum of zero to a maximum score of 100. A score of 91-100 is excellent, 81-90 is good, 71-80 is fair, 70 or below is poor. The patient records the following: pain level, need for assistance when walking, presence of a limp, distance able to walk, ability to put on shoes and socks, climb stairs, use public transportation and the length of time one is able to comfortably sit in a chair are all scored.
Time Frame: The Harris Hip Total Score evaluation took place at 6 weeks, 6 months, 12 months, and a final evaluation at 24 months or greater (up to 96 months)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System | Pinnacle™ Acetabular Cup With Marathon® Polyethylene
Number analyzed (Participants) | 177 | 87
Units on a scale
  Pre-operative | 50.5 (9.6) | 50.8 (9.5)
  6 weeks | 75.7 (12.3) | 73.6 (12.7)
  6 months | 92.2 (11.4) | 91.4 (11.6)
  12 months | 94.2 (10.1) | 93.7 (9.6)
  last follow up of 24 months or greater | 94.6 (9.3) | 94.5 (8.0)
Statistical Analysis 1: Comparison: Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System vs Pinnacle™ Acetabular Cup With Marathon® Polyethylene; Test type: Non-Inferiority or Equivalence — This was a non-inferiority test of the Harris Hip Score means at 24+ months with a 5 point non-inferiority margin; p = 0.001, ANCOVA; Preoperative Harris Hip score was included in the ANCOVA model as the only covariate; Mean Difference (Final Values) = 0.61, 95% CI 1-sided [lower limit -1.56]

2. Secondary Outcome: Complication Rates
Description: Complication Rates are reported by each type of complication (adverse events/AEs) in the Adverse Events Tab
Time Frame: The Complication Rates were evaluated at 6 weeks, 6 months, 12 months, and a final evaluation at 24 months or greater (up to 96 months)
Population: Complication Rates are contained in the Adverse Events Tab and include all reported complications in all patients as represented in the Final Clinical Study Report
Measure: Number; unit: Complications
Groups:
- Investigational; Control: Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System The Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup Prosthesis System consists of a modular ceramic bearing insert that attaches to a Pinnacle™ Acetabular Shell by a taper locking mechanism. The ceramic insert is designed to articulate against a 28 mm ceramic femoral head that is attached to a conventional femoral stem to complete the total hip prosthesis.
Arm/Group | Investigational | Control
Number analyzed (Participants) | 177 | 87
Complications | 567 | 287

ADVERSE EVENTS:
Arm/Group | Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System | Pinnacle™ Acetabular Cup With Marathon® Polyethylene
All-Cause Mortality (participants affected / at risk) | 4/177 | 3/87
Serious Adverse Events (participants affected / at risk) | 27/177 | 14/87
Other Adverse Events (participants affected / at risk) | 80/177 | 44/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System (N=177) | Pinnacle™ Acetabular Cup With Marathon® Polyethylene (N=87)
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Endocrine/Metabolic (Endocrine disorders) | 1 (1) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 16 (16) | 8 (8)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Neurological (Nervous system disorders) | 1 (1) | 0 (0)
Genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acetabular liner failure (Surgical and medical procedures) | 1 (1) | 0 (0)
Femoral Component Loosening (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delta Ceramax™ Ceramic-on-Ceramic Acetabular Cup System (N=177) | Pinnacle™ Acetabular Cup With Marathon® Polyethylene (N=87)
Cardiovascular (Cardiac disorders) | 11 (11) | 6 (6)
Wound Problem (Injury, poisoning and procedural complications) | 9 (9) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 68 (68) | 36 (36)
Genitourinary (Renal and urinary disorders) | 10 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.